CLINICAL TRIAL: NCT05897749
Title: Clinical Study on the Effect of Brucea Javanica Oil Emulsion Injection on the Survival of Patients With Advanced Colorectal Cancer Who Failed to Receive Multi-line Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ying Zhang, professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZYYCXTD-C-202205
Record Dates: First submitted 2023-05-09; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Chinese Herbal Medicine; Progression-free Survival; Quality of Life
Keywords: Colorectal Cancer; Javanica oil emulsion injection; Chinese Herbal Medicine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Brucea javanica oil emulsion injection+The best supportive treatment (Experimental)
  Interventions: Other: Brucea javanica oil emulsion injection; Other: The best supportive treatment
- control group:The best supportive treatment (Active Comparator)
  Interventions: Other: The best supportive treatment

INTERVENTIONS:
Other: Brucea javanica oil emulsion injection — Drug: Brucea javanica oil emulsion injection Brucea javanica oil emulsion injection: intravenous drip, 30ml each time (add 250ml sterile physiological saline),once a day, 14 consecutive days as a cycle, at least 2 cycles completed. The best supportive treatment:According to the NCCN Best Palliative Treatment Guidelines (2022. V1), provide the best supportive treatment
  Arms: Experimental group: Brucea javanica oil emulsion injection+The best supportive treatment
Other: The best supportive treatment — The best supportive treatment:According to the NCCN Best Palliative Treatment Guidelines (2022. V1), provide the best supportive treatment

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of Brucea javanica oil emulsion injection in patients with advanced colorectal cancer who failed to undergo multi-line treatment

DETAILED DESCRIPTION:
this study included a prospective, multicenter, randomized controlled clinical trial.

About 60 patients will be recruited in the randomized clinical trial. Participants will be randomly divided into experimental group (n=30) and control group (n=30). The patients in the experimental group will receive Brucea javanica oil emulsion injection combined with the best supportive treatment, based on the NCCN best palliative treatment guidelines (2022. V1). The patients in the control group received the best supportive treatment based on the NCCN's best palliative treatment guidelines (2022. V1). The primary end point was PFS (progression-free survival). The research protocol was approved by the relevant ethics committee. The research was conducted in accordance with the Helsinki Declaration and good clinical practice guidelines. The patient has written informed consent to participate in the trial.

ELIGIBILITY:
Inclusion Criteria:

* # Colorectal cancer patients with stage IV third line or above treatment failure confirmed by pathology

  * Male or female aged 18-75years # Eastern Cooperative Oncology Group (ECOG) performance score 0-2
  * Life expectancy of at least 3 months # At least one radiographically measurable lesion per RECIST 1.1 # Willing to join the clinic trail and sign informed consent,and able to comply with scheduled visits and treatments

Exclusion Criteria:

* With brain metastasis, BRAF-V600E mutation, HER-2 overexpression, MSI-H, NTRK fusion gene patients

  * Patients with primary tumors at other sites
  * Pregnant or breastfeeding woman
  * Fertile patients who are unwilling or unable to take effective contraceptive measures during the research period until 6 months after the study end later
  * A history of mental disorders # Patients with severe cardiac, cerebrovascular, liver, kidney, hematopoietic system dysfunction or primary disease without effective control # Participated in other clinical trials of small molecule research drugs within 28 days prior to enrollment, or participated in other clinical trials of large molecule research drugs within 3 months before enrollment # Known allergy or intolerance to study medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-16 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Randomization until disease progression, death, or 12 months after randomized enrollment, whichever occurs first.]
  Progression Free Survival

SECONDARY OUTCOMES:
ORR | Every two cycles(each cycle is 28 days) until disease progression, death, or 12 months after randomized enrollment, whichever occurs first.
  Objective Response Rate
quality of life | Before and after each cycle (each cycle is 28 days) of treatment, assessed up to 12 months after randomized enrollment, equlity of life assessed by the MDASI. The higher the score, the worse the quality of life.
  equlity of life assessed by the MDASI [followed by its scale information in the Description]")
quality of life | Before and after each cycle (each cycle is 28 days) of treatment, assessed up to 12 months after randomized enrollment, equlity of life assessed by the EORTC QLQ-C30. The higher the score, the worse the quality of life.
  equlity of life assessed by the EORTC QLQ-C30 [followed by its scale information in the Description]")

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu, China
  - The Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong, China
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine,Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be issued to publications through scientific journals and conference reports.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Fang L, Wang Y, Fang Y, Wang R, Xie Y, Yang S, Liu S, Zhang Y. Brucea javanica oil emulsion plus supportive care for refractory advanced colorectal cancer: a pilot RCT protocol. Front Pharmacol. 2025 Jul 21;16:1610575. doi: 10.3389/fphar.2025.1610575. eCollection 2025. PMID 40761400